CLINICAL TRIAL: NCT05252910
Title: Collection of Specimens From Adult and Adolescent Participants ≥12 Years Old Who Will Receive an Authorized or Licensed COVID-19 Vaccine as Part of Usual Care
Brief Title: Specimen Collection Study From Coronavirus Disease 2019 (COVID-19) Vaccinated Adults and Adolescents
Acronym: CoVacSpec
Status: Terminated | Type: Observational
Why Stopped: Global spread of SARS-CoV-2 Omicron variant and vaccination preclude ability to enroll sufficient SARS-CoV-2 seronegative participants.
Sponsor: Pharm-Olam, LLC (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2021SPEC-001
Record Dates: First submitted 2022-02-10; First posted 2022-02-23 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Coronavirus Disease 2019 (COVID-19); Specimen collection; Severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, peripheral blood mononuclear cells, serum, RNA, DNA, and nasal mucosa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a specimen collection study intended to generate a biological specimen repository of samples from severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) naïve adults and adolescents ≥12 years old who will receive locally authorized or licensed COVID-19 vaccines. Approximately 1,000 participants will be enrolled.

Plasma and peripheral blood mononuclear cell samples will be obtained either by venipuncture, or by leukapheresis. Serum, RNA, and DNA samples will be obtained by venipuncture. Specimens for mucosal antibody assessments will be collected by nasal swabbing.

Biological specimens will be collected from study participants at Baseline prior to the COVID-19 vaccine dose and at timepoints aligned with the study participant's vaccination schedule for a period of up to 1 year following receipt of the initial COVID-19 vaccination.

DETAILED DESCRIPTION:
This specimen collection study will generate a bank of biological specimens/samples and associated meta data from severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2) naïve adults and adolescent participants ≥12 years old who will receive authorized or licensed Coronavirus Disease 2019 (COVID-19) vaccine as a matter of care. The samples may be used to determine immunological responses and microbiologic factors, to develop novel assays, diagnostic tests, therapeutic agents, and vaccines.

Vaccines received by study participants will be only those supported and approved for use by the United States Government, and authorized or licensed for use in the country in which the participant is enrolled. Participants will be receiving COVID-19 vaccine as a matter of standard preventive medical care, and not as a research activity. Participant screening and biological specimen collection will occur only after informed consent/assent. Participants may participate in all, or a part, of this study to provide biological specimens.

Participants who are eligible for the study will be stratified into age groups: ≥12 to <18 years, ≥18 to ≤65 years, >65 years of age. Approximately 1,000 participants will be enrolled in this study.

Biological specimens will be collected from each participant for up to 1 year following receipt of their initial COVID-19 vaccination. Additional participants may be enrolled for up to 2 additional years.

Enrollment dynamics will be actively monitored across all sites, and efforts will be made to balance enrollment by sex, age group, and type of vaccine received. Testing of blood samples obtained from study participants at screening will be performed on an ongoing basis to assess for evidence of prior COVID-19 infection. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) serostatus of participants across the program will be actively monitored to target an enrollment of at least 75% seronegative participants for both adult as well as adolescent participants.

Demographic data, height and weight, vaccination details, major past medical history, and comorbidities will be collected at baseline from study participants. Concomitant medications, significant intercurrent medical events, and unanticipated adverse events or problems posing risks to study subjects will be recorded from enrollment through the end of the study for all participants.

There is no analysis plan or primary or secondary endpoints for this specimen collection study. The study will be conducted in accordance with Good Clinical Practices for human research solely for the purpose of generating a repository of serial blood (collected by phlebotomy and leukapheresis) and nasal swab specimens from severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2) naïve adults and adolescents ≥12 years old who have received authorized or licensed COVID-19 vaccines.

Samples will be identified only by subject identification number.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant (by participant report) female adults (≥18 years or older) or adolescents (≥12 years old and <18 years old) in generally good health, who will receive a locally licensed or authorized COVID-19 vaccine, development of which was supported by the United States Government, as part of standard preventive medical care.
* Able to understand and sign the Informed Consent Form (for adolescent participants informed consent form from parent and participant assent).
* Participants with some medical conditions that might otherwise disqualify them from routine blood or blood component donations, such as HIV/AIDS, diabetes mellitus, etc., can participate if their conditions are stable, well-controlled, have had no change in clinical status or medication for at least 6 months, and whose participation in the protocol would not present excess risk to the participant as judged by the Investigator.
* Willing to comply with study procedures and schedule for sample collections.
* Available for follow-up visits over the next year.

For individuals willing to undergo leukapheresis procedure(s), Adults ≥18 years, and adolescents ≥12-17 years must meet the following minimum criteria:

* Weight ≥110 pounds/50 kg
* Platelet count >150×109/L
* Adequate bilateral antecubital veins to allow for 2 peripheral vein access points.
* At least 2 weeks since any previous blood product donation.

Exclusion Criteria:

* Prior receipt of any COVID-19 vaccine.
* Anemia at screening, or history of anemia caused by chronic therapies or congenital/genetic conditions (e.g., thalassemia) per participant/parent report. Individuals with histories of anemias that have been remedied with treatment (e.g., parasitism, B12, iron deficiency) are allowed.
* Have a history of intravenous drug abuse.
* Have a history of sickle cell disease per participant/parent report
* Have a history of poorly controlled or clinically significant heart, lung, kidney disease, per participant/parent report and Investigator assessment.
* Have a history of Hepatitis B or C, per participant/parent report. Participants with resolved Hepatitis B or C, or those with no apparent clinical manifestations of these infections, may participate.
* Have a contraindication to phlebotomy (i.e., evidence of cellulitis or abscess; venous thrombosis on palpation; presence of hematoma; presence of vascular shunt, graft, or access device; anti-coagulation therapy; history of bleeding diathesis; or clinically significant thrombocytopenia (platelet count <150×109/L) as assessed by Investigator, participant/parent report, or screening platelet count.
* Have a history of untreated, unresolved, or recurrent malaria during the preceding 12 months per participant/parent report.
* Have donated blood in the past 8 weeks.
* Have planned surgery in the next 8 weeks.
* Is breast feeding, pregnant, or may be pregnant, per participant report.
* Are currently participating or are planning to participate in any clinical trial, including a COVID-19 vaccine trial or COVID-19 therapeutic trial.
* Any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study.
* Any condition that in the judgement of the Investigator precludes participation because it could adversely affect participant safety or data integrity.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males or non-pregnant (by participant report) females
Study Population: The study population will consist of subjects meeting the inclusion/exclusion criteria who are SARS-CoV-2 naïve adults and adolescents ≥12 years old who will receive locally authorized or licensed COVID-19 vaccines. All subjects must be willing to assent/sign the informed consent and undergo venipuncture, nasal swab collection, and leukapheresis (where allowed and subject agrees).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Specimen Collection | 12 months (1 year)
  This study is designed to collect biological specimens/samples to generate a biological specimen repository of samples from severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2) naïve adults and adolescent participants ≥12 years old who will be receiving, as a matter of care, locally authorized or licensed Coronavirus Disease 2019 (COVID-19) vaccines whose development has been supported by the US Government. Specimens collected with associated metadata will be shared with the US Government and stakeholders.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly McKee, MD, Principal Investigator — Pharm-Olam, LLC
Locations (32):
- United States (6):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - SUNY Upstate Medical University, Syracuse, New York
  - Meharry Medical College/Meharry Medical Center, Nashville, Tennessee
  - Pan American Clinical Research LLC, Brownsville, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
- Colombia (3):
  - Clinisalud, Envigado, Antioquia
  - Bluecare Salud SAS, Bogotá, Columbia
  - Servimed SAS, Bucaramanga, Santander Department
- University Hospital Center of Guadeloupe, Les Abymes, Guadeloupe
- India (7):
  - Andhra Medical College, Visakhapatnam, Andhra Pradesh
  - Unity Hospital, Surat, Gujarat
  - GMERS Medical College & Hospital, Vadodara, Gujarat
  - Government Medical College & Hospital, Aurangabad, Maharashtra
  - Govt. Medical College, Nagpur, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Peerless Hospitex Hospital, Kolkata, West Bengal
- Icaro Investigaciones en Medicina SA de CV, Chihuahua City, Mexico
- CAIMED Center at the Ponce School of Medicine, Ponce, Puerto Rico
- South Africa (13):
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - REIMED Wilhase Practice, Boksburg, Gauteng
  - Clinresco Centres, Kempton Park, Gauteng
  - Larisha Pillay-Ramaya, Pretoria, Gauteng
  - Muhammed Ameen Fulat, Pretoria, Gauteng
  - Johan Geldenhuys, Vereeniging, Gauteng
  - DR P J Sebastian Clinical Research Centre, Durban, KwaZulu-Natal
  - Synapta Clinical Research Centre, Durban, KwaZulu-Natal
  - Clinical Research Institute of South Africa (CRISA), KwaDukuza, KwaZulu-Natal
  - Aurum Klerksdorp CRS, Klerksdorp, North West
  - The Aurum Institute, Rustenburg Clinical Research Site, Rustenburg, North West
  - Langeberg Clinical Trials, Cape Town, Western Cape
  - Task Applied Science, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No